CLINICAL TRIAL: NCT05761002
Title: Human Papilloma Virus Genotypes and Treatment Outcomes of Intralesional Immunotherapy of Anogenital Warts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Rana Ehab, lecturer of dermatology, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 94412022
Record Dates: First submitted 2023-02-26; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Human Papilloma Virus; Anogenital Wart
MeSH Terms: conditions — Condylomata Acuminata | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): All patients will be subjected to:
  * A thorough history taking and proper dermatological examination.
  * Skin sampling from anogenital wart lesions: skin sterilization followed by injection of local anesthesia at the base of lesions, then the part of wart above skin surface will be removed using shave biopsy technique.
  * DNA extraction of skin samples.
  * Conventional PCR for low-risk HPV genotypes (6,11) and RT-PCR for high-risk HPV genotypes.
  * Intralesional injection of the quadrivalent HPV vaccine (Gardasil) at a dose of 0.5ml, into the largest wart at 4-week intervals until complete clearance is achieved or for a maximum of three sessions.
  Interventions: Biological: the Quadrivalent Vaccine (Gardasil)

INTERVENTIONS:
Biological: the Quadrivalent Vaccine (Gardasil) — • Intralesional injection of the quadrivalent HPV vaccine (Gardasil) at a dose of 0.5ml, into the largest wart at 4-week intervals until complete clearance is achieved or for a maximum of three sessions.

SUMMARY:
This study aims to investigate the relationship between HPV genotypes and treatment outcomes of intralesional immunotherapy of anogenital warts with the quadrivalent vaccine (Gardasil).

DETAILED DESCRIPTION:
Human papillomavirus (HPV), a member of the Papillomaviridae family, is a small, icosahedral, non-enveloped virus with a circular double-stranded DNA genome. Sexually transmitted HPV, which mainly infects mucosal and keratinized epithelium, has a cytopathic effect on the epithelium. Genital mucosal HPV infection is persistent and multifocal and can be subclinical (Alacam & Bakir, 2021). Infection with HPV causes a large proportion of cervical, vaginal, vulvar, anal, and penile cancers, as well as genital warts (Choi, 2019).

Anogenital warts are common benign dermatological conditions caused by different HPV genotypes, with serotypes 6, 11, 16, and 18 being the most causative types (Santos-López et al., 2015). Their prevalence varies according to geographical locations. Data is not yet available on the HPV burden in the general population of Egypt (Elazab et al., 2021). In October 2014, a very important multicenter observational study in Egypt concluded that the prevalence of HPV among Egyptian women aged 18 years or more is about 10.4%, with the highest prevalence of HPV infection being observed among women aged 45-54 years (Shaltout et al., 2014).

Different modalities are available for the treatment of warts, such as topical podophyllin, imiquimod, podophyllotoxin, or trichloroacetic acid, surgical excision, electrosurgery, cryosurgery, laser surgery, and intralesional immunotherapy (Gill, 2021; Nofal et al., 2022). Available treatments are time-consuming, painful, and can leave scars or hypopigmentation. Furthermore, recurrence rates after any treatment range from 6% to 100% (Ciccarese et al., 2019). As a result, there has been a demand for safer modalities to treat recalcitrant warts. Immunotherapy presents an alternative approach to the management of warts as it provides ease of application, but even distant lesions get resolved with application to a single lesion. Immunotherapy has been performed with imiquimod, BCG vaccine, HPV vaccines, and auto implantation therapy (Gill, 2021).

Three HPV vaccines are licensed as protective measures against the development of genital warts, cervical cancer, and other anogenital cancers. They include the bivalent vaccine targeting serotypes 16/18 (Cervarix), the quadrivalent vaccine targeting serotypes 6/11/16/18 (Gardasil), and the nonavalent vaccine targeting serotypes 6/11/16/18/31/33/45/52/58 (Gardasil-9) (Vaccine Information Statement | HPV | VIS | CDC, 2021). There is a strong immune response against the HPV vaccine that not only causes the clearance of local wart lesions but also causes the clearance of distant lesions. The vaccine is designed to elicit neutralizing antibody responses which prevent initial infection with HPV, but in warts it mainly acts by mounting cell-mediated and humoral responses which help in the clearance of warts. The quadrivalent HPV vaccine contains inactive L1 proteins from four different strains: 6, 11, 16, and 18; synthesized in the yeast Saccharomyces cerevisiae (Gill, 2021).

ELIGIBILITY:
Inclusion Criteria:

- Patients with clinically diagnosed multiple anogenital warts who had not received treatment in the last 2 months before the study

Exclusion Criteria:

* Patient refusal, pregnancy, lactation, age less than 10 years, and immunosuppressive conditions

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
improvement of lesion | 6 month
  The response will be considered complete if there is disappearance of the warts, partial if the warts regressed in size by 50-99% and no response if there is 0-49% decrease in wart size.

CONTACTS AND LOCATIONS:
Locations (1):
- Rana Ehab, Zagazig, Egypt